CLINICAL TRIAL: NCT03096990
Title: An Observational Study of the Real-life Management of Psoriatic Arthritis Patients Treated With Otezla® (Apremilast) in Belgium
Brief Title: A Study of the Real-life Management of Psoriatic Arthritis Patients Treated With Otezla® (Apremilast) in Belgium
Acronym: APOLO
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004-PSA-010; U1111-1194-0305 (Other: UTN Number)
Record Dates: First submitted 2017-03-24; First posted 2017-03-31 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic Arthritis; Observational; Otezla; Apremilast; Real-Life management; Belgium; APOLO; CC-10004
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Use of apremilast in patients with active PsA: Psoriatic arthritis patients treated with Otezla® (apremilast) in Belgium
  Interventions: Drug: apremilast

INTERVENTIONS:
Drug: apremilast — Psoriatic arthritis patients treated with Otezla® (apremilast) in Belgium

SUMMARY:
The study will include a representative sample of 150 patients with active Psoriatic Arthritis (PsA) for whom the treating rheumatologist has decided to begin treatment with apremilast. This study is non-interventional, drug dosing and treatment duration will be at the sole discretion of the treating rheumatologist, in accordance with the local label and daily clinical practice. APOLO is a national (Belgium), multicentre, prospective, non-interventional, post-marketing study.

DETAILED DESCRIPTION:
Patient care will follow routine clinical practice, involving regular follow-up visits, without any mandatory visit. In daily practice, patients are usually seen by their treating rheumatologist every 3 months. In this study, patients will be followed-up for a least 6 months and at most 18 months after apremilast treatment initiation. Patient data will be collected until 31st December 2018. Assuming a recruitment phase of 18-month duration starting as of December 2016, individual patient follow-up times will range from 6 to 18 months, depending on the inclusion date. During the first months of the study, the recruitment rate has been slower than expected. Therefore, it has been decided in October 2017 to increase the period of recruitment to 18 months in order to have enough evaluable patients to keep the accuracy required for the statistical analysis.

During the study, it is expected to collect data at inclusion and at 6 months after apremilast initiation in all patients. As per NIHDI recommendations, patients should consult their treating rheumatologists 6 months after apremilast initiation in order to evaluate treatment response and decide on treatment continuation for an additional period of 12 months. For patients recruited early in the study, data will be collected during the next follow-up visits up to 18 months after apremilast initiation. Only data pertaining to visits occurring at 9 (± 1), 12 (± 1), 15 (±1), and 18 (± 1) months after treatment initiation will be collected. If a study visit occurs approximately 3 (± 1) months after treatment initiation, the data will also be recorded.

All clinical data collected during this non-interventional study will be routinely documented in the patient's medical records, which are the main source of information. The study data will be collecting via an electronic Case Report Form (eCRF). Data from source documents including PRO-questionnaires will be entered in the eCRF by the investigator or other authorised appropriately designed and trained study site personnel. Data entered into the eCRF will be reviewed for consistency by the Data Manager using both automated logical checks (issuing in automatic queries generated by the system) and manual review (issuing in manual checks set by the Data Manager or the Monitor into the eCRF). All data collected within the eCRF will be approved and electronically signed and dated by the Investigator or designee. At the conclusion of the study, before the final statistical analysis, the eCRF and other study data will be locked to further additions or corrections.

During the study, the Clinical Research Associate (CRA) will contact each study site on a regular basis in order to check the progress and conduct of the study. If issues regarding study conduct arise, additional on-site visits may be performed. In particular, a quality analysis will also be performed and based on data quality, it will be decided whether on-site monitoring is necessary, for which site and on which percentage of patients. During monitoring visits, eCRFs, patient's source documents, and all other study documentation will be reviewed by the CRA. Accuracy will be checked by performing source data verification that is a direct comparison of the entries made onto the eCRF against the appropriate source documentation.

Adverse events AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) terminology.

The detailed methodology of the statistical analyses will be documented in a statistical analysis plan (SAP). The SAP will be written by the Clinical Research Organisation (CRO) in charge of the study and will be validated by sponsor prior to performing the analysis and obligatory before the database lock. A scientific committee has been selected for this study. This committee will provide advice on the SAP.

ELIGIBILITY:
Inclusion Criteria:

- Patients who meet ALL the following criteria can be enrolled:

* Male or female aged at least 18 years,
* With a diagnosis of active Psoriatic Arthritis (PsA),
* For whom the treating physician has made the decision to commence apremilast treatment in accordance with the local label and reimbursement criteria (refer to the reimbursement conditions mentioned in Section 1.2),
* Able to follow the instructions of the study,
* Having signed an Informed Consent Form (ICF).

Exclusion Criteria:

- Patients who meet AT LEAST one of the following exclusion criteria will be excluded:

* Women who are pregnant, breastfeeding or planning on becoming pregnant,
* Non-menopausal women who are not using an adequate contraception method,
* Patients with hypersensitivity to apremilast or to one of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with active PsA visiting rheumatology practices in Belgium and eligible for treatment with apremilast according to the local label and reimbursement criteria. The decision to treat the patient with apremilast will be made prior to the decision to enter the patient into the study.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing response assessed by improvement for at least 2 out of 4 measures which compose the Psoriatic Arthritis Response Criteria (PsARC) at 6 months after apremilast initiation with respect to baseline | 6 months after Apremilast initiation
  The PsARC tool is a composite response measure that has been specifically developed to assess response to treatment in Psoriatic Arthritis (PsA). PsARC is considered as an acceptable primary endpoint by the European Medicines Agency (EMA) The response for a given subject is defined by an improvement for at least 2 out of 4 measures which compose the PsARC (Patient Global Assessment [PtGA] of disease activity, Patient Global Assessment [PGA] of disease activity, 68-joint count for pain/tenderness and 66 joint count for swelling) and no worsening in any of the 4 measures.

SECONDARY OUTCOMES:
Characteristics of the patients treated with apremilast | Baseline
  The patients treated with Apremilast will be described according to the following characteristics: demographics (age, gender, weight, height, and ethnicity), professional status, lifestyle habits, medical history (including psoriasis and PsA treatment
Change from baseline in measures which compose the PsARC (PtGA of disease activity, PGA of disease activity, 68-joint count for pain/tenderness, and 66-joint count for swelling) | up to 18 months
  The PsARC tool is a composite response measure that has been specifically developed to assess response to treatment in PsA. PsARC is considered as an acceptable primary endpoint by the European Medicines Agency (EMA) The response for a given subject is defined by an improvement for at least 2 out of 4 measures which compose the PsARC (Patient Global Assessment [PtGA] of disease activity, Patient Global Assessment [PGA] of disease activity, 68-joint count for pain/tenderness and 66 joint count for swelling) and no worsening in any of the 4 measures.
Change from Baseline in Psoriatic Arthritis Impact Of Disease 12 [PsAID12] score | up to 18 months
  The total score is divided by 20 and the final score ranges from 0 to 10, where '10' represents the worst health score. PsAID 12 is a questionnaire assessing 12 domains (pain, fatigue, skin, work and/or leisure activities, function, discomfort, sleep, coping, anxiety, embarrassment, social life, and depression) based on a 0-10 NRS, each parameter having a different coefficient.
Change from Baseline in Health Assessment Questionnaire Disability Index [HAQ-DI] score | up to 18 months
  The Health Assessment Questionnaire (HAQ) is a validated PRO questionnaire designed to measure health status and health-related quality of life. It consists of 20 items covering activities of daily living classified in 8 domains. Respondents indicate for every item whether they can do the activity 'without any difficulty', with 'some' or 'much difficulty' or are 'unable to do' the activity. The HAQ yields a disability index (HAQ-DI) score between 0 and 3, where, 0 means no functional disability and 3 represents severe functional disability.
Change from Baseline in disease activity Numerical Rating Scale (NRS) | up to 18 months
  Is an 11-point horizontal scale anchored at 0 and 10, with 0 representing "no disease activity" and 10 representing "maximal disease activity".
  The patient's global self-assessment of disease activity is measured on a 0 to 10 unit NRS. The physician's global assessment of disease activity is also measured on a 0 to 10 unit NRS. For patient's assessment and for the physician's assessment, the NRS
Change from Baseline in pain/itch Visual Analogue Scale [VAS] | up to 18 months
  The patient is asked to mark the line at the point that best represented the intensity of his or her pain and itch respectively. The VAS numeric values are the distances in millimeters from "no pain" and "no itch" respectively to the points marked by the patient. The pain VAS consists of a 100-mm horizontal line anchored at one end with the words "no pain" and at the other end with the words "worst possible pain".
Change from Baseline in body surface area (BSA) | up to 18 months
  The investigator evaluates the percentage involvement of psoriasis on each participant's BSA on a continuous scale from 0% = no involvement to 100% = full involvement, where 1% corresponded to the size of the participant's handprint including the palm, fingers, and thumb
Change from Baseline in Leeds Enthesitis Index (LEI) | up to 18 months
  The LEI was developed specifically for use in PsA. It measures enthesitis at 6 sites (lateral epicondyle, left and right; medial femoral condyle, left and right; Achilles tendon insertion, left and right). Each site is assigned a score of 0 (absent) or 1 (present); the results from each site is then added to produce a total score (range 0 to 6).
Change from Baseline in Dactylitis score | up to 18 months
  Each digit on the hands and feet is rated as zero for no dactylitis or 1 for dactylitis present. The dactylitis severity score is the sum of the individual scores for each digit. The dactylitis severity score, ranging from 0 to 20, is the number of digits on the hands and feet with dactylitis present. Dactylitis is characterized by swelling of the entire finger or toe.
Mean duration of treatment with apremilast in biologic-naïve patients and in patients having received a previous biological treatment. | up to 18 months
  Time to the stop of the treatment by Apremilast will be calculated as the time interval from the date of apremilast initiation to the date of the apremilast stop
Rate and reasons for discontinuation of apremilast treatment within 6 months after initiation | Up to 6 months
  Descriptive statistics will be provided for the rate and reasons for discontinuation of treatment within 6 months. This analysis will be performed on safety population and restricted to patients who stop the treatment before the time point to analyse or for which the follow-up is at least so long as the time point to analyse.
Adverse Events (AEs) | up to 18 months
  Number of participants with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (22):
- Belgium (22):
  - ASZ Aalst, Aalst
  - Onze Lieve Vrouw Aalst, Aalst
  - AZ Sint-Jan, Bruges
  - CHU St Pierre (César de Paepe), Brussels
  - Clinicque Saint-Jean Botanique, Brussels
  - CHU Brugmann, Brussels
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - Cliniques Universiatires Saint-Luc, Brussels
  - Private Practice, Céroux-Mousty
  - UZ Antwerpen, Edegem
  - Reumacentrum Genk, Genk
  - Reumaclinic, Genk
  - UZ Gent, Ghent
  - GHdC Site Saint-Joseph, Gilly
  - CHU UCL Mont-Godinne, Godinne
  - Reuma Instituut, Hasselt
  - AZ Zeno campus Knokke-Heist, Knokke-Heist
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
  - Reumatologie Medizorg, Merksem
  - ZNA Jan Palfijn, Merksem
  - Private Practice, Uccle

REFERENCES:
- [Derived] de Vlam K, Toukap AN, Kaiser MJ, Vanhoof J, Remans P, Van den Berghe M, Di Romana S, Van den Bosch F, Lories R. Real-World Efficacy and Safety of Apremilast in Belgian Patients with Psoriatic Arthritis: Results from the Prospective Observational APOLO Study. Adv Ther. 2022 Feb;39(2):1055-1067. doi: 10.1007/s12325-021-02016-x. Epub 2022 Jan 3. PMID 34977986
- See also: Expanded Access for CC-10004 — https://clinicaltrials.gov/ct2/show/NCT03096990?term=CC-10004-PSA-010&rank=1